CLINICAL TRIAL: NCT00922051
Title: Acute Effects of Acu-TENS on FEV1 and Blood β-Endorphin Level in Subjects With COPD
Brief Title: Acute Effects of Acu-Transcutaneous Electrical Nerve Stimulation (Acu-TENS) on Forced Expiratory Flow Volume in One Second (FEV1) and Blood β-Endorphin Level in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice Jones, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSEARS20070305001
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; FEV1; beta endorphin; TENS; acupuncture
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Application of Acu-TENS
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Group 2 (Placebo Comparator)
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS)
  Arms: Group 1
Device: Transcutaneous electrical nerve stimulation (TENS) — Placebo
  Arms: Group 2

SUMMARY:
The objective of this study is to investigate the effectiveness of Acu-TENS (transcutaneous electrical nerve stimulation applied on acupoints) on lung functions, dyspnoeic symptoms and its association with beta endorphin level in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis with COPD

Exclusion Criteria:

* allergic to gel
* unable to perform spirometry
* unable to communicate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Forced expiratory flow volume in one second (FEV1), forced vital capacity (FVC) | measured before and after intervention

SECONDARY OUTCOMES:
Beta endorphin | before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alice Jones, PhD, FACP, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China